CLINICAL TRIAL: NCT01902017
Title: Randomized, Double Blind, Placebo Controlled Trial of Ketotifen in Patients With Elbow Fractures or Dislocations
Brief Title: Investigations of Mechanisms and Treatment in Post-traumatic Joint Contractures
Acronym: Ketotifen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); American Society for Surgery of the Hand (Other); Workers' Compensation Board, Alberta (Other)
Responsible Party: Principal Investigator, Dr. Kevin Hildebrand, Orthopaedic Surgeon, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REB15-0081; REB15-0081 (Other: Conjoint Health Research Ethics Board)
Record Dates: First submitted 2013-07-10; First posted 2013-07-17 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Joint Contractures
Keywords: Joint; Contracture; Elbow; Fracture; Dislocation
MeSH Terms: conditions — Contracture; Fractures, Bone; Joint Dislocations | interventions — Ketotifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Operative, Ketotifen (Experimental): Ketotifen 5mg orally twice per day for 6 weeks.
  Interventions: Drug: Ketotifen
- Non-operative, Ketotifen (Experimental): Ketotifen 5mg orally twice per day for 6 weeks.
  Interventions: Drug: Ketotifen
- Operative, Placebo (Placebo Comparator): Placebo oral medication twice daily for 6 weeks.
  Interventions: Drug: Placebo
- Non-operative, Placebo (Placebo Comparator): Placebo oral medication twice daily for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketotifen — 5 mg PO bid
  Other Names: Zaditen
  Arms: Non-operative, Ketotifen; Operative, Ketotifen
Drug: Placebo — 5 mg placebo PO bid
  Other Names: Lactose Placebo
  Arms: Non-operative, Placebo; Operative, Placebo

SUMMARY:
Injured joints, especially at the elbow, are at risk for permanent motion loss, also known as joint contractures. Joint contractures limit the function of an elbow and are a recognized complication that occurs often after a traumatic injury. The benefits of early motion after injury has helped in preventing joint contractures but there are still several patients that develop debilitating joint contractures. Current research suggests that mast cells, which are found in the joint, are key in causing joint contractures. Research has been done using a medication called Ketotifen. Ketotifen has been linked to stabilizing mast cells and preventing the joint contracture. It is hoped that short-term use of this medication after an injury will prevent the contracture from occurring.

DETAILED DESCRIPTION:
Individuals ≥ 18 years old with isolated distal 1/3 humerus and/or proximal 1/3 ulna and/or proximal 1/3 radius fractures and/or elbow dislocations (open fractures with or without nerve injury may be included) and presented to Peter Lougheed Centre (PLC), Foothills Medical Center (FMC), or South Health Campus (SHC).

Participants were required to take Ketotifen 5mg by mouth twice a day for 6 weeks or placebo twice a day by mouth for 6 weeks. Neither the participant nor the physician knew if the participant was taking Ketotifen or placebo. Sometimes this type of injury requires surgery. This study invited both patients that do and do not require surgery to participate.

We took a sample of blood to measure tryptase (normally found in the body). We predicted people with high levels of tryptase were more likely to develop stiffening in the joint.

Participants were asked to return for follow up visits 2, 6, 12, 24, and 52 weeks after surgery or date of initial injury if surgery was not required. These visits were part of normal care for this type of injury.

At the visit participants were asked to do the following, some of which was not part of normal care.

At each visit: Range of motion of the elbow was assessed, DASH score was completed- form helping the research group understand the level of disability from this injury, X-rays until the fracture was considered healed (this was normal treatment), SF12 - questionnaire about how the patient was feeling and coping with their injury, Additional information was collected about how the injury was healing and weight was measured.

The participant was required to have physiotherapy which is normal treatment for this injury.

The participant was contacted by telephone at week 1, 3, 4 and 5 while taking the study medication. During these times:

The participant was asked about:

* any problems with the study medication
* any new conditions or concerns that have developed

The participant was reminded:

* of next visit
* to continue to take study drug as instructed

During these telephone contacts, if any problems were detected that could not be rectified or figured out during the telephone interview, then participant was asked to attend the Cast Clinic to see their doctor in person.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Isolated distal 1/3 humerus fractures
* Proximal 1/3 ulna fractures
* Proximal 1/3 radial fractures
* Elbow dislocations
* Open fractures with or without nerve injury
* Presentation to Peter Lougheed Centre (PLC), Foothills Medical Centre (FMC) or South Health Campus (SHC).

Exclusion Criteria:

* Pre-existing elbow contracture
* Osteoarthritis of affected elbow
* Inflammatory arthritis of affected elbow
* Gout of affected elbow
* Nonspecific monoarticular arthritis of the affected elbow
* Inability to give informed consent due to irreversible cognitive disorder
* Inability to comply with post-operative physiotherapy
* Injury > 7 days at the time of presentation
* Inability to mobilize elbow injury within 2 weeks of injury or surgery
* Pregnancy
* Breast feeding
* Oral hypoglycemic medications
* History of epilepsy
* Lactose intolerance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-06; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Joint range of motion | 12 months post-injury
  Extension-flexion arc of motion

SECONDARY OUTCOMES:
Range of motion | 2,6,12,24 and 52 weeks post injury
Patients requiring (re)operation for elbow-related causes | 12 months
Radiographic evaluation for fracture healing/non-union | 12-52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Hildebrand, MD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - Peter Lougheed Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta

REFERENCES:
- [Background] Liu CS, Ademola A, Zhang M, Garven A, Kopka M, Salo PT, Hart DA, Befus AD, Hildebrand KA. Human serum mast cell tryptase levels in elbow fractures or dislocations and its association with injury severity. J Orthop Res. 2020 Sep;38(9):2015-2019. doi: 10.1002/jor.24642. Epub 2020 Mar 11. PMID 32112583
- [Derived] Hildebrand KA, Schneider PS, Mohtadi NGH, Ademola A, White NJ, Garven A, Walker REA, Sajobi TT; PERK 1 Investigators. PrEvention of Posttraumatic contractuRes with Ketotifen 1 (PERK 1): A Randomized Clinical Trial. J Orthop Trauma. 2020 Dec 1;34(12):e442-e448. doi: 10.1097/BOT.0000000000001878. PMID 32639394